CLINICAL TRIAL: NCT03420781
Title: A 46-week, Double-blind, Placebo-controlled, Phase 3 Study With a 6-week Randomized-withdrawal Period to Evaluate the Safety and Efficacy of Relamorelin in Patients With Diabetic Gastroparesis
Brief Title: A Safety and Efficacy Study of Relamorelin in Diabetic Gastroparesis Study 03
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Relamorelin program is being terminated solely based on a business decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLM-MD-03
Record Dates: First submitted 2018-01-24; First posted 2018-02-05 (Actual); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: diabetic gastroparesis; vomiting
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus; Vomiting | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Period: Placebo (Placebo Comparator): Placebo-matching relamorelin injected subcutaneously twice daily for up to 40 weeks.
  Interventions: Drug: Placebo
- Treatment Period: Relamorelin 10 μg (Experimental): Relamorelin 10 micrograms (μg) injected subcutaneously twice daily for up to 40 weeks.
  Interventions: Drug: Relamorelin
- Randomized Withdrawal Period: Placebo then Relamorelin 10 μg (Experimental): Participants who received placebo-matching relamorelin injected subcutaneously twice daily for 40 weeks, followed by relamorelin 10 μg injected twice daily for up to 6 weeks in the Randomized Withdrawal (RW) Period.
  Interventions: Drug: Placebo; Drug: Relamorelin
- Randomized Withdrawal Period: Relamorelin 10 μg then Relamorelin 10 μg (Experimental): Participants who received relamorelin 10 μg injected subcutaneously twice daily for 40 weeks, followed by relamorelin injected twice daily for up to 6 weeks in the RW Period.
  Interventions: Drug: Relamorelin
- Randomized Withdrawal Period: Relamorelin 10 μg then Placebo (Experimental): Participants who received relamorelin 10 μg injected subcutaneously twice daily for 40 weeks, followed by placebo-matching relamorelin injected twice daily for up to 6 weeks in the RW Period.
  Interventions: Drug: Placebo; Drug: Relamorelin

INTERVENTIONS:
Drug: Placebo — Placebo injected twice daily
  Arms: Randomized Withdrawal Period: Placebo then Relamorelin 10 μg; Randomized Withdrawal Period: Relamorelin 10 μg then Placebo; Treatment Period: Placebo
Drug: Relamorelin — Relamorelin 10 μg injected twice daily
  Arms: Randomized Withdrawal Period: Placebo then Relamorelin 10 μg; Randomized Withdrawal Period: Relamorelin 10 μg then Placebo; Randomized Withdrawal Period: Relamorelin 10 μg then Relamorelin 10 μg; Treatment Period: Relamorelin 10 μg

SUMMARY:
A 46-week study to compare the efficacy of relamorelin with that of placebo in participants with diabetic gastroparesis (DG). At the end of the 40-week Treatment Period, participants will either continue on relamorelin or placebo for 6 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all the following criteria apply:
* Participant met all inclusion/exclusion criteria of either Protocol RLM-MD-01 (NCT03285308) or Protocol RLM-MD-02 (NCT03426345) and successfully completed the study
* Able to provide written informed consent (IC) prior to any study procedures and willing and able to comply with study procedures
* In the opinion of the investigator, the participant demonstrated adequate compliance with the study procedures in Study RLM-MD-01 or RLM-MD-02

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Participant is not willing or able to abide by the restrictions regarding concomitant medicine use
* Participant is planning to receive an investigational drug (other than study treatment) or investigational device at any time during Study RLM-MD-03
* Participant has an unresolved adverse event (AE) or a clinically significant finding on physical examination, clinical laboratory test, or 12-lead electrocardiogram (ECG) that, in the investigator's opinion, would limit the participant's ability to participate in or complete the study
* Any other reason that, in the investigator's opinion, would confound proper interpretation of the study or expose a participant to unacceptable risk, including renal, hepatic or cardiopulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw Bochenek, Study Director — Allergan
Locations (337):
- United States (161):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Digestive Health Specialist of the South East, Dothan, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Del Sol Research Management, LLC, Chandler, Arizona
  - Phoenix Clinical LLC., Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Unity Health - Searcy Medical Center, Searcy, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Aurora Care Clinic, LLC, Costa Mesa, California
  - Diagnamics Inc., Encinitas, California
  - VVCRD Research, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Angel City Research Inc., Los Angeles, California
  - TriWest Research Associates, Poway, California
  - Medical Associates Research Group, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Upland Clinical Research, Upland, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Synexus Clinical Research US, Inc. - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Gastroenterology Associates of Fairfield County, P.C., Bridgeport, Connecticut
  - TrialSpark, Inc., Washington D.C., District of Columbia
  - Innovative Research of West FL, Inc., Clearwater, Florida
  - West Central Gastroenterology, Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - ALL Medical Research LLC, Cooper City, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - Vida Clinical Trials, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - APF Research LLC, Miami, Florida
  - AMPM Research Clinic, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - American Research Institute, Inc, Miami, Florida
  - Panax Clinical Research, LLC., Miami Lakes, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Synexus, Pinellas Park, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gwinnett Research Institute, LLC, Buford, Georgia
  - Summit Clinical Research, LLC., Carnesville, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - Clinical Research Consultants of Atlanta, Suwanee, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Research, LLC, Jeffersonville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Health Science Research Center, Pratt, Kansas
  - WestGlen Gastrointestinal Consultants, Shawnee Mission, Kansas
  - Cotton-O'Neil Clinical Research Center - Digestive Health, Topeka, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Via Christi Clinic, PA, Wichita, Kansas
  - Tri-State Gastroenterology, Crestview Hills, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - WK Physicians Network, Bossier City, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Cronola LLC, Houma, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - New Orleans Research Institute - Metropolitan Gastroenterology Associates, Metairie, Louisiana
  - Clinical Trials of America, Inc., West Monroe, Louisiana
  - Trialspark - Silverman, Bowie, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Frederick Gastroenterology Associates, PA an Elligo Health Research Site, Frederick, Maryland
  - Woodholme Gastroenterology Associates, P.A., Glen Burnie, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Commonwealth Clinical Studies, PLLC., Brockton, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Vida Clinical Studies, Dearborn, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Minnesota Gastroenterology, P.A., Coon Rapids, Minnesota
  - Montana Medical Research, Missoula, Montana
  - Methodist Physicians Clinic Diabetes and Endocrine Specialists, Omaha, Nebraska
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Garden State Endocrinology, Brick, New Jersey
  - AGA Clinical Research Associates LLC, Egg Harbor, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Synexus Clinical Research US, Inc., Jamaica, New York
  - United Health Services Hospitals, Inc., Johnson City, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolina Digestive Health Associates, PA, Concord, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Vidant Multispeciality Clinic - Kinston, Kinston, North Carolina
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - PMG Research Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Diabetes & Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Synexus Clinical Research US - Cincinnati, Cincinnati, Ohio
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - CIC America Clinical Inquest Center Ltd., Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Premier Clinical Research d.b.a. STAT Research, Franklin, Ohio
  - Family Practice Center of Wadsworth, Inc. DBA New Venture Medical Research, Wadsworth, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Family Medical Associates, Research Department, Levittown, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Synexus Clinical Research US, Inc, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinsearch, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Avant Research Associates,LLC, Austin, Texas
  - ClinRx Research, LLC, Carrollton, Texas
  - Synexus Clinical Research US, Inc., Dallas, Texas
  - Biopharma Informatic Inc., Research Center, Houston, Texas
  - Rodriguez Clinical Trials, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - Advanced Research Institute, Inc., Ogden, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Verity Research Inc., Fairfax, Virginia
  - Manassas Clinical Research Centre, Manassas, Virginia
  - Cardinal Internal Medicine Associates, PC, Woodbridge, Virginia
  - Washington Gastroenterology PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (9):
  - Maffei Centro Medico-Investigacion Clinica Aplicada, C.a.b.a., Buenos Aires
  - Hospital Sirio Libanes, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Privado de Investigaciones Clínicas de Córdoba, Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas de Rosario, Rosario, Santa Fe Province
  - Instituto de Hematologia y Medicina Clinica Dr. Ruben Davoli, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - CIPREC, Buenos Aires
  - Centro Universitario de Investigacion en Farmacologia Clinic, Corrientes
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (4):
  - Ordination, Sankt Stefan ob Stainz, Styria
  - VIVIT Institute, am LKH Feldkirch, Feldkirch, Vorarlberg
  - Privatklinik Wehrle-Diakonissen, Salzburg
  - Landeskrankenhaus Steyr, Steyr
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Gastro-Enterologie,, Edegem, Antwerp
  - UZ Brussel, Jette, Brussels Capital
  - AZ Sint Lucas Brugge, Bruges, West-Vlaanderen
- Brazil (10):
  - Instituto de Estudos e Pesquisas Clinicas do Ceará IEP/CE - Oncology, Fortaleza, Ceará
  - Hospital Universitário Walter Cantídio, Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto Catarinense de Endocrinologia e Diabetes (ICED), Joinville, Santa Catarina
  - Scentryphar Pesquisa Clinica Ltda, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - CPQuali Pesquisa Clinica Ltda, Santa Cecília, São Paulo
  - Hospital Universitário João de Barros Barreto, Belém
  - IPEC-Instituto de Pesquisa Clinica, São Paulo
- Bulgaria (2):
  - MHAT Yuliya Vrevska Byala, Byala, Ruse
  - UMHAT - Kaspela- EOOD, Plovdiv
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Central Alberta Research Centre, Red Deer, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Recherche GCP Research, Montreal, Quebec
- Colombia (11):
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Centro Cardiovascular Colombiano Clínica Santa María, Medellín, Antioquia
  - Centro Cardiovascular y de Diabetes, Barranquilla, Atlántico
  - Fundacion BIOS, Barranquilla, Atlántico
  - Medplus Medicina Prepagada, Bogotá, Bogota D.C.
  - Asociación Colombiana de Diabetes, Teusaquillo, Bogota D.C.
  - Endocare Ltda., Bogotá, Cundinamarca
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Fundacion Centro de Investigaciones Clinicas CARDIOMET, Pereira, Risaralda Department
  - Centro Medico Imbanaco de Cali S.A., Cali, Valle del Cauca Department
  - IPS Centro Medico Julian Coronel S.A, Cali, Valle del Cauca Department
- Denmark (2):
  - Gentofte Hospital, Hellerup, Copenhagen
  - Gastroenheden, Hvidovre hospital, Hvidovre, Copenhagen
- Germany (6):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - Studienzentrum Schwittay, Böhlen, Saxony
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Clinical Research Hamburg, Hamburg
  - Israelitisches Krankenhaus, Hamburg
  - KRH Klinikum Siloah, Hanover
- Hungary (6):
  - First Department of Medicine, University of Szeged, Szeged, CsonfrÃ¡d
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger, Heves County
  - Hetenyi Geza Hospital, Tószeg, Jász-Nagykun-Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg, Zala County
  - Synexus Budapest DRS, Budapest
  - Strázsahegy Gyógyszertár Medicina, Budapest
- India (21):
  - Kumudini Devi Diabetes Research Center; Ramdevrao Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Dr. Jivraj Mehta Smarak Health Foundation, Bakeri Medical Research Centre, Ahmedabad, Gujarat
  - Victoria Hospital, Bangalore, Karnataka
  - Life Care Hospital & Research Centre, Bangalore, Karnataka
  - Diacon Hospital and research Center - Diabetology, Bengaluru, Karnataka
  - Rajalakshmi Hospital, Bengaluru, Karnataka
  - Vinaya Hospital & Research Centre, Mangalore, Karnataka
  - Bhatia Hospital, Mumbai, Maharashtra
  - B. J. Government Medical College and Sassoon General Hospitals, Pune, Maharashtra
  - Universal Hospital, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - S.R. Kalla (SRK) Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Diabetic Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - Eternal Hospital - Diabetology, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Kovai Diabetes Speciality Centre, Coimbatore, Tamil Nadu
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - M. V Hospital & Research Centre, Lucknow, Uttar Prandesh
  - Sir Ganga Ram Hospital, New Delhi
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Endocrinology & Diabetes Center, Safed
- Latvia (4):
  - Kraslava Hospital, Krāslava, Kraslavas Nov.
  - Polana-D, Daugavpils
  - Pauls Stradins Clinical University Hospital, Endokrinologijas nodala, Riga
  - Digestive Diseases Centre GASTRO, Riga
- Malaysia (3):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Universiti Sains Malaysia, Kubang Kerian
  - Hospital Taiping, Taiping
- Mexico (13):
  - Centro de Investigación y Atención de Diabetes - Endocrinología y Nutrición, Durango, Guillermina
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente, S.C., Guadalajara, Jalisco
  - Consultorio Medico, Guadalajara, Jalisco
  - Unidad de Investigación Clínica en Medicina S.C., Guadalajara, Jalisco
  - Mentrials SA DE CV, Cuauhtémoc, Mexico City
  - Clinicos Asociados BOCM SC, Mexico City, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevencion de E - Endocrinology, Mexico City, Mexico City
  - Centro de Atención e Investigación en Factores de Riesgo Car, México, Mexico DF
  - Centro de Desarrollo Biomédico S.C.P, Mérida, Yucatán
  - Centro de Investigacion Cardiometabolica de Aguascalientes SA de CV, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Dioderm Instituto de Investigacion, Durango
  - Sociedad de Metabolismo y Corazon, S.C., Veracruz
- Philippines (7):
  - West Visayas State University Medical Center, Iloilo City, IloIlo
  - Manila Doctors Hospital, Ermita, Manila, Metropolitan Manila
  - San Juan De Dios Educational Foundation, Inc., Pasay, Metropolitan Manila
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Cardinal Santos Medical Center, San Juan City, National Capital Region
  - Ospital ng Makati, Makati City, NCR
  - Perpetual Succor Hospital, Cebu City
- Poland (5):
  - NZOZ Vita Diabetica - Malgorzata Buraczyk, Bialystok, Podlaski
  - Endoskopia Sp. Z O.O., Sopot, Pomeranian Voivodeship
  - Centrum Medyczne Lukamed, Chojnice
  - Specjalistyczny Gabinet Neurologiczny Marta Banach, Krakow
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
- Russia (11):
  - Saint-Petersburg City Pokrovskaya Hospital, St-Petersburg, Leningradskaya Oblast'
  - Scientific Institute of Clinical and Experimental Lymphology, Novosibirsk, Novosibirsk Oblast
  - North-Western State Medical University named after I. I. Mechnikov, Saint Petersburg, Sankt-Peterburg
  - Nizhegorodsky Regional Clinical Hospital named after N. A. Semashko, Nizhny Novgorod, Volga
  - Kazan State Medical University, Kazan'
  - FSBI National medical endocrinology research centre, Moscow
  - Moscow Regional Research Clinical Institute named by MF Vladimirski, Moscow
  - Rostov on Don, Rostov-on-Don
  - Rostov State Medical University, Rostov-on-Don
  - GUZ Saratov City Clinical Hospital 9, Saratov
  - Saratov City Clinical Hospital 12, Saratov
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (5):
  - FARMOVS, Bloemfontein, Free State
  - Wits Clinical Research, Johannesburg, Gauteng
  - Synexus Stanza Clincal Reaserch Centre, Pretoria, Gauteng
  - Watermeyer Clinical Research Site, Pretoria, Gauteng
  - Synexus Helderberg Clinical Research Centre, Cape Town, Western Cape
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Diabetes Center, Seoul, Nowon-gu
  - Asan Medical Center, Seoul
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Ukraine (22):
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Regional muniRegional municipal institution "Chernivtsi's regional clinical hospital", gastroenterological department, Higher state educational establishment of Ukraine "Bukovinian state medical university", department of internal medicine and infectious, Chernivtsi
  - Regional Public Organization "Chernivtsi Regional Endocrinology Center", Chernivtsi
  - State Institution Ukrainian State Research Institute of Medical and Social Problems of Disability of the Ministry of Health of Ukraine, Dnipro
  - Municipal nonprofit entity of Kharkiv municipal council, Kharkiv
  - L.T.Malaya Therapy National Institute of the National Academy of Medical Sciences of Ukraine, Kharkiv
  - Clinical Endocrinology of SI "V.Danilevsky Institute for endocrine pathology problems National Academy of Medical sciences of Ukraine", Kharkiv
  - Communal Institution Kherson City Clinical Hospital, Kherson
  - Limited Liability Company "Medical and Diagnostic Center "ADONIS Plus", outpatient department, c. Kyiv, Kyiv
  - Kyiv clinical hospital on railway transport #2 of the "Healthcare Centre" branch of JSC "Ukrainian Railway", Kyiv
  - Medical Center Universal Clinic Oberig, Kyiv
  - Polyclinic of medical services and rehabilitation department of State Joint-Stock Holding Company Artem, day-patient unit, Kyiv
  - Odessa Railway Clinical Hospital of Branch of HC JSC Ukrzaliznytsia, Odessa National Medical University, Odesa
  - Communal Institution "Odesa Regional Clinical Hospital", Out-patient department, Odesa
  - Poltava Regional Clinical Hospital, Poltava
  - Ternopil University Hospital, Ternopil
  - Private Small-Scale Enterprise Medical Centre Pulse, Vinnytsia
  - Vinnytsia Regional Clinical highly specialized Endocrinology Centre, Vinnytsia
  - Municipal nonprofit entity "Vinnytsia's city clinical hospital #1", c. Vinnytsia, Vinnytsia
  - 6th City Clinical Hospital, c. Zaporizhzhia, Zaporizhzhia
  - Municipal Institution, City Hospital #7, Zaporizhzhia
- United Kingdom (10):
  - Biomedical Research Centre, Nottingham, East Midland
  - MAC Clinical Research Manchester, Manchester, Greater Manchester
  - Royal Oldham Hospital, Oldham, Lancashire
  - MAC Research, Exchange House, Cannock, Staffordshire
  - MAC Clinical Research, Monarch House, Leeds, West Yorkshire
  - MAC Research, Barnsley
  - MAC Clinical Research, Kaman Court, Blackpool
  - Mid Essex Hospital Services NHS Trust Broomfield Hospital, Chelmsford
  - MAC Clinical Research, Liverpool
  - MAC Clinical Research, GAC House, Stockton-on-Tees

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed RLM-MD-01 [NCT03285308] or RLM-MD-02 [NCT03426345] were eligible for enrollment.
Period: Treatment Period (40 Weeks)
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Started | 236 | 231 | 0 | 0 | 0
Safety Population (Safety Population included all participants in the Intent-to-treat (ITT) population who received ≥1 administration of study treatment.) | 235 | 231 | 0 | 0 | 0
Completed (Out of 197 participants who completed the Treatment Period, 193 entered the RW Period.) | 92 | 105 | 0 | 0 | 0
Not Completed | 144 | 126 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 6 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 16 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 6 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 2 | 0 | 0 | 0
Not completed — Study Terminated by the Sponsor | 101 | 89 | 0 | 0 | 0
Not completed — Site Terminated by the Sponsor | 1 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 3 | 0 | 0 | 0 | 0
Period: RW Period: 6 Weeks (Week 41 to Week 46)
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Started | 0 | 0 | 91 | 59 | 43
Completed | 0 | 0 | 85 | 54 | 38
Not Completed | 0 | 0 | 6 | 5 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Study Terminated by the Sponsor | 0 | 0 | 6 | 3 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population included all participants who entered the 40-week treatment period.
Groups:
- Treatment Period: Relamorelin 10 μg: Relamorelin 10 μg injected subcutaneously twice daily for up to 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Total
Number analyzed (Participants) | 236 | 231 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.11) | 56.2 (11.51) | 55.9 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 166 | 328
  Male | 74 | 65 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 82 | 165
  Not Hispanic or Latino | 153 | 149 | 302
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 8 | 11
  Asian | 21 | 18 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 21 | 58
  White | 175 | 183 | 358
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Diabetic Gastroparesis Symptom Severity Score (DGSSS) of the Treatment Period
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the Diabetic Gastroparesis Symptom Severity Diary (DGSSD), recorded in an electronic diary (e-diary). The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to Week 12 of this study
Population: Modified-intent-to-treat (mITT) Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
score on a scale
  Baseline | 24.9 (5.65) | 24.8 (6.28)
  Change from Baseline to Week 12: number analyzed (Participants) | 205 | 202
  Change from Baseline to Week 12 | -11.9 (9.43) | -11.2 (9.00)

2. Primary Outcome: Percentage of Participants Meeting the Vomiting Responder Criterion During Each of the Last 6 Weeks of the First 12-weeks of the Treatment Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. A Vomiting Responder was defined as a participant with zero weekly vomiting episodes during each of the last 6 weeks of the first 12-weeks of the 40-week Treatment Period.
Time Frame: Week 6 to Week 12
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 29.4 | 21.4

3. Secondary Outcome: Percentage of Participants Meeting the Nausea Responder Criterion During Each of the Last 6 Weeks of the First 12-weeks of the Treatment Period
Description: A Nausea Responder was defined as a participant with improvement (decrease) of at least 2-points in the weekly symptom scores for nausea at each of the last 6 weeks of the first 12-weeks of the 40-week Treatment Period. Nausea was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0=no nausea to 10=worst possible nausea. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 6 to Week 12)
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 46.0 | 43.2

4. Secondary Outcome: Percentage of Participants Meeting the Abdominal Pain Responder Criterion During Each of the Last 6 Weeks of the First 12-weeks of the Treatment Period
Description: An Abdominal Pain Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for abdominal pain at each of the last 6 weeks of the first 12-weeks of the 40-week Treatment Period. Abdominal pain was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0=no abdominal pain to 10=the worst possible abdominal pain and was recorded in an e-diary. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 6 to Week 12)
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 40.4 | 39.7

5. Secondary Outcome: Percentage of Participants Meeting the Bloating Responder Criterion During Each of the Last 6 Weeks of the First 12-weeks of the Treatment Period
Description: A Bloating Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for bloating at each of the last 6 weeks of the first 12-weeks of the 40-week Treatment Period. Bloating was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0=no bloating and 10=the worst possible bloating and was recorded in the e-diary. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 6 to Week 12)
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 38.3 | 38.4

6. Secondary Outcome: Percentage of Participants Meeting the Postprandial Fullness Responder Criterion During Each of the Last 6 Weeks of the First 12-weeks of the Treatment Period
Description: A Postprandial Fullness Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for Postprandial Fullness at each of the last 6 weeks of the first 12-weeks of the 40-week Treatment Period. Postprandial Fullness was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0=no feeling of fullness until finishing a meal (best) to 10=feeling full after only a few bites (worst). Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 6 to Week 12)
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 36.6 | 36.2

7. Secondary Outcome: Change From Baseline to Week 40 in the Average Weekly DGSSS of the Treatment Period
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the DGSSD, recorded in an e-diary. The DGSSS was derived as the sum of the weekly averages (Week 37 to Week 40) of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period of the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 37 to Week 40)
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
score on a scale
  Baseline | 24.9 (5.65) | 24.8 (6.28)
  Change from Baseline to Week 40: number analyzed (Participants) | 112 | 123
  Change from Baseline to Week 40 | -13.3 (10.22) | -12.3 (9.20)

8. Secondary Outcome: Percentage of Participants Meeting the Vomiting Responder Criterion at Week 40 of the Treatment Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. A Vomiting Responder was defined as a participant with zero weekly vomiting episodes during the last 4 weeks of the 40-week Treatment Period.
Time Frame: Week 37 to Week 40
Population: mITT Population included all participants in the ITT population with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
percentage of participants | 19.1 | 18.8

9. Secondary Outcome: Change From Baseline to Week 40 in the Average Weekly Number of Vomiting Episodes of the Treatment Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. The average weekly number of vomiting episodes were derived as the average of the weekly number of vomiting episodes in the last 4 weeks of the 40-week Treatment Period. A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 37 to Week 40)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: vomiting episodes per week
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 235 | 229
vomiting episodes per week
  Baseline | 6.8 (11.09) | 7.3 (11.52)
  Change from Baseline to Week 40: number analyzed (Participants) | 112 | 123
  Change from Baseline to Week 40 | -1.8 (17.51) | -5.4 (11.87)

10. Secondary Outcome: Change From Baseline to Week 46 in the Average Weekly DGSSS of the Randomized-Withdrawal Period
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the DGSSD, recorded in an e-diary. The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). Average weekly scores are derived as the average of the weekly scores from the 6 weeks of the RW Period. A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 41 to Week 46)
Population: RW Population included all participants who were re-randomized or assigned to a treatment of RW Period and received ≥1 administration of study treatment during the RW Period. Overall number analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg: Participants who received placebo-matching relamorelin injected subcutaneously twice daily for 40 weeks, followed by relamorelin 10 μg injected twice daily for up to 6 weeks in the RW Period.
Arm/Group | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 91 | 58 | 43
score on a scale
  Baseline | 25.7 (5.65) | 25.7 (6.25) | 24.4 (5.47)
  Change from Baseline to Week 46: number analyzed (Participants) | 86 | 56 | 39
  Change from Baseline to Week 46 | -13.4 (10.45) | -12.5 (9.71) | -12.5 (9.35)

11. Secondary Outcome: Change From Baseline to Week 46 in the Average Weekly Number of Vomiting Episodes of the Randomized-Withdrawal Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. Average weekly number of vomiting episodes are derived as the average of the weekly number of vomiting episodes from the six weeks of the RW Period. A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period in the previous studies.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02) to (Week 41 to Week 46)
Population: RW Population included all participants who were re-randomized or assigned to a treatment of RW Period and received ≥1 administration of study treatment during the RW Period. Overall number analyzed are the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: vomiting episodes per week
Arm/Group | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 91 | 58 | 43
vomiting episodes per week
  Baseline | 6.1 (7.01) | 9.9 (11.92) | 4.2 (4.73)
  Change from Baseline to Week 46: number analyzed (Participants) | 86 | 56 | 39
  Change from Baseline to Week 46 | -1.8 (18.40) | -7.3 (10.23) | -1.8 (6.12)

12. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is an AE that begins or worsens after receiving study drug.
Time Frame: First dose of study drug to within 30 days of the last dose of study drug (Up to approximately 50 weeks)
Population: Safety Population included all participants in the ITT population who received ≥1 administration of study treatment in Treatment Period. RW Population included all participants who were re-randomized or assigned to a treatment of RW population and received ≥1 administration of study treatment during the RW Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 235 | 231 | 91 | 59 | 43
Participants | 129 | 131 | 18 | 12 | 8

13. Secondary Outcome: Number of Participants With Potential Clinically Significant (PCS) Clinical Laboratory Results
Description: Clinical Laboratory values included Hematology, Chemistry and Urinalysis tests. The investigator determined if the results were clinically significant. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to 46 weeks
Population: Safety Population included all participants in the ITT population who received ≥1 administration of study treatment in Treatment Period. RW Population included all participants who were re-randomized or assigned to a treatment of RW population and received ≥1 administration of study treatment during the RW Period. Number analyzed is the number of participants with non-PCS Baseline values and at least one postbaseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 235 | 231 | 91 | 59 | 43
Participants
  Eosinophils Absolute Cell Count [10^9/liter(L)]: >3×Upper Limit of Normal Value (ULN): number analyzed (Participants) | 227 | 225 | 91 | 59 | 43
  Eosinophils Absolute Cell Count [10^9/liter(L)]: >3×Upper Limit of Normal Value (ULN) | 2 | 1 | 0 | 1 | 1
  Hematocrit (RATIO): >1.1×ULN: number analyzed (Participants) | 214 | 224 | 86 | 59 | 42
  Hematocrit (RATIO): >1.1×ULN | 1 | 2 | 2 | 1 | 0
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN): number analyzed (Participants) | 214 | 224 | 86 | 59 | 42
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN) | 7 | 7 | 4 | 0 | 2
  Hemoglobin [grams (g)/L]: <0.9×LLN: number analyzed (Participants) | 214 | 220 | 86 | 58 | 42
  Hemoglobin [grams (g)/L]: <0.9×LLN | 13 | 14 | 5 | 1 | 4
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 226 | 221 | 90 | 57 | 42
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN | 1 | 4 | 0 | 0 | 0
  Mean Corpuscular Volume [femtoliter (fL)]: >1.1×ULN: number analyzed (Participants) | 222 | 224 | 89 | 59 | 43
  Mean Corpuscular Volume [femtoliter (fL)]: >1.1×ULN | 2 | 3 | 1 | 0 | 0
  Mean Corpuscular Volume (fL): <0.9×LLN: number analyzed (Participants) | 222 | 224 | 89 | 59 | 43
  Mean Corpuscular Volume (fL): <0.9×LLN | 4 | 0 | 1 | 0 | 0
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 224 | 221 | 90 | 57 | 41
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN | 0 | 2 | 2 | 0 | 0
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 224 | 221 | 90 | 57 | 41
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN | 6 | 4 | 2 | 0 | 0
  Platelet Count (Thrombocytes) (10^9/L): >1.5×ULN: number analyzed (Participants) | 227 | 224 | 91 | 59 | 42
  Platelet Count (Thrombocytes) (10^9/L): >1.5×ULN | 0 | 1 | 0 | 0 | 0
  Platelet Count (Thrombocytes) (10^9/L): <0.5×LLN: number analyzed (Participants) | 227 | 224 | 91 | 59 | 42
  Platelet Count (Thrombocytes) (10^9/L): <0.5×LLN | 1 | 0 | 0 | 0 | 0
  Red Blood Cell Count (10^12/L): >1.1×ULN: number analyzed (Participants) | 223 | 224 | 90 | 58 | 42
  Red Blood Cell Count (10^12/L): >1.1×ULN | 1 | 0 | 0 | 0 | 0
  Red Blood Cell Count (10^12/L): <0.9×LLN: number analyzed (Participants) | 223 | 224 | 90 | 58 | 42
  Red Blood Cell Count (10^12/L): <0.9×LLN | 4 | 8 | 4 | 1 | 0
  White Blood Cell Count (10^9/L): <0.7×LLN: number analyzed (Participants) | 227 | 225 | 91 | 59 | 42
  White Blood Cell Count (10^9/L): <0.7×LLN | 2 | 0 | 0 | 0 | 0
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN: number analyzed (Participants) | 227 | 225 | 91 | 59 | 43
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN | 2 | 2 | 0 | 2 | 1
  Albumin (g/L): <0.9×LLN: number analyzed (Participants) | 225 | 226 | 90 | 59 | 43
  Albumin (g/L): <0.9×LLN | 1 | 1 | 1 | 0 | 1
  Alkaline Phosphatase (U/L): >=3×ULN: number analyzed (Participants) | 227 | 226 | 91 | 59 | 43
  Alkaline Phosphatase (U/L): >=3×ULN | 0 | 3 | 0 | 0 | 0
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN: number analyzed (Participants) | 227 | 225 | 91 | 59 | 42
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN | 3 | 2 | 0 | 0 | 0
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN: number analyzed (Participants) | 223 | 218 | 91 | 58 | 41
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN | 3 | 2 | 1 | 1 | 0
  Bicarbonate (HCO3) (mmol)/L: >0.9×LLN: number analyzed (Participants) | 223 | 218 | 91 | 58 | 41
  Bicarbonate (HCO3) (mmol)/L: >0.9×LLN | 6 | 9 | 2 | 4 | 1
  Bilirubin, Total [micromoles(μmol)/L]: >1.5×ULN: number analyzed (Participants) | 227 | 226 | 91 | 59 | 43
  Bilirubin, Total [micromoles(μmol)/L]: >1.5×ULN | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): >1.2×ULN: number analyzed (Participants) | 207 | 207 | 84 | 52 | 39
  Blood Urea Nitrogen (mmol/L): >1.2×ULN | 29 | 20 | 8 | 4 | 4
  Calcium (mmol/L): >1.1×ULN: number analyzed (Participants) | 225 | 221 | 90 | 57 | 42
  Calcium (mmol/L): >1.1×ULN | 1 | 0 | 1 | 0 | 0
  Calcium (mmol/L): <0.9×LLN: number analyzed (Participants) | 225 | 221 | 90 | 57 | 42
  Calcium (mmol/L): <0.9×LLN | 1 | 0 | 0 | 0 | 1
  Chloride (mmol/L): <0.9×LLN: number analyzed (Participants) | 227 | 226 | 91 | 59 | 43
  Chloride (mmol/L): <0.9×LLN | 2 | 1 | 1 | 0 | 1
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN: number analyzed (Participants) | 221 | 222 | 90 | 59 | 43
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN | 4 | 1 | 0 | 1 | 0
  Creatinine (μmol/L): >1.3×ULN: number analyzed (Participants) | 211 | 213 | 84 | 51 | 41
  Creatinine (μmol/L): >1.3×ULN | 22 | 16 | 5 | 2 | 3
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN: number analyzed (Participants) | 206 | 201 | 84 | 56 | 41
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN | 41 | 33 | 9 | 9 | 4
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN: number analyzed (Participants) | 206 | 201 | 84 | 56 | 41
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN | 14 | 9 | 4 | 2 | 2
  Glycohemoglobin A1C: Increase of >=0.5%: number analyzed (Participants) | 224 | 223 | 91 | 59 | 43
  Glycohemoglobin A1C: Increase of >=0.5% | 134 | 138 | 62 | 26 | 28
  Glycohemoglobin A1C: Increase of >=1%: number analyzed (Participants) | 224 | 223 | 91 | 59 | 43
  Glycohemoglobin A1C: Increase of >=1% | 134 | 138 | 62 | 26 | 28
  Phosphorus (mmol/L): >1.1×ULN: number analyzed (Participants) | 221 | 219 | 88 | 56 | 43
  Phosphorus (mmol/L): >1.1×ULN | 10 | 12 | 4 | 4 | 4
  Phosphorus (mmol/L): <0.9×LLN: number analyzed (Participants) | 221 | 219 | 88 | 56 | 43
  Phosphorus (mmol/L): <0.9×LLN | 4 | 3 | 0 | 0 | 0
  Potassium (mmol/L): <0.9×LLN: number analyzed (Participants) | 227 | 226 | 91 | 59 | 43
  Potassium (mmol/L): <0.9×LLN | 0 | 0 | 2 | 0 | 0
  Protein, Total (g/L): >1.1×ULN: number analyzed (Participants) | 225 | 226 | 90 | 59 | 43
  Protein, Total (g/L): >1.1×ULN | 0 | 1 | 0 | 0 | 0
  Protein, Total (g/L): <0.9×LLN: number analyzed (Participants) | 225 | 226 | 90 | 59 | 43
  Protein, Total (g/L): <0.9×LLN | 0 | 1 | 0 | 0 | 1
  Triglycerides, Fasting (mmol/L): >=3×ULN: number analyzed (Participants) | 217 | 216 | 87 | 58 | 42
  Triglycerides, Fasting (mmol/L): >=3×ULN | 9 | 11 | 4 | 4 | 2
  Uric Acid (Urate) (μmol/L): >1.1×ULN: number analyzed (Participants) | 192 | 181 | 77 | 44 | 35
  Uric Acid (Urate) (μmol/L): >1.1×ULN | 31 | 31 | 5 | 3 | 1
  Uric Acid (Urate) (μmol/L): <0.9×LLN: number analyzed (Participants) | 192 | 181 | 77 | 44 | 35
  Uric Acid (Urate) (μmol/L): <0.9×LLN | 3 | 4 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Meaningful Trends for Vital Signs
Description: Vital Signs included assessments of heart rate, respiratory rate, systolic and diastolic blood pressure, and body temperature. The investigator determined if the results were clinically significant.
Time Frame: Up to 46 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 235 | 231 | 91 | 59 | 43
Participants | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results
Description: A standard 12-lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 46 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 235 | 231 | 91 | 59 | 43
Participants | 3 | 2 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With a ≥1% Increase in Glycosylated Hemoglobin A1c (HBA1c)
Time Frame: Up to 46 weeks
Population: Safety Population included all participants in the ITT population who received ≥1 administration of study treatment in Treatment Period. RW Population included all participants who were re-randomized or assigned to a treatment of RW population and received ≥1 administration of study treatment during the RW Period. Overall number analyzed is the number of participants with non-PCS Baseline values and at least one postbaseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
Number analyzed (Participants) | 224 | 223 | 91 | 59 | 43
Participants | 134 | 138 | 62 | 26 | 28

17. Secondary Outcome: Number of Participants With Anti-relamorelin Antibody Testing Results
Description: A blood sample was collected that was sent to a laboratory for an anti-relamorelin antibody screening test. A positive screening test was confirmed by an immunodepletion assay.
Time Frame: Up to 46 weeks
Population: Due to limitations at the vendor's end, the final analysis data could not be obtained.
Arm/Group | Treatment Period: Relamorelin 10 μg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of the last dose of study drug (Up to approximately 50 weeks)
Description: All-Cause Mortality: all randomized participants. Adverse Events: Safety Population included all participants in the ITT population who received ≥1 administration of study treatment in Treatment Period; RW Population included all participants who were re-randomized or assigned to a treatment of RW population and received ≥1 administration of study treatment during the RW Period.
Arm/Group | Treatment Period: Placebo | Treatment Period: Relamorelin 10 μg | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo
All-Cause Mortality (participants affected / at risk) | 3/236 | 2/231 | 0/91 | 0/59 | 0/43
Serious Adverse Events (participants affected / at risk) | 24/235 | 20/231 | 3/91 | 2/59 | 1/43
Other Adverse Events (participants affected / at risk) | 18/235 | 27/231 | 0/91 | 0/59 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Placebo (N=235) | Treatment Period: Relamorelin 10 μg (N=231) | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg (N=91) | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg (N=59) | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo (N=43)
Coronary artery disease (Cardiac disorders) | 3 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Postinfarction angina (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychogenic tremor (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 3 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Placebo (N=235) | Treatment Period: Relamorelin 10 μg (N=231) | Randomized Withdrawal Period: Placebo Then Relamorelin 10 μg (N=91) | Randomized Withdrawal Period: Relamorelin 10 μg Then Relamorelin 10 μg (N=59) | Randomized Withdrawal Period: Relamorelin 10 μg Then Placebo (N=43)
Urinary tract infection (Infections and infestations) | 13 | 16 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 12 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03420781/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03420781/SAP_001.pdf